CLINICAL TRIAL: NCT02447523
Title: The Impact of Metabolic Syndrome on Patients Undergoing Elective Laparotomy
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Petros Tzimas, Assistant Professor of Anaesthesiology, University of Ioannina
Other Study IDs: 19/17-10-2012
Record Dates: First submitted 2015-05-05; First posted 2015-05-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Metabolic Syndrome; Anesthesia; Perioperative Outcome; Complications
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with metabolic syndrome: Patients fulfilling criteria to establish the diagnosis of metabolic syndrome
  Interventions: Procedure: Elective abdominal surgery
- Patients without metabolic syndrome: Patients not fulfilling criteria of the metabolic syndrome
  Interventions: Procedure: Elective abdominal surgery

INTERVENTIONS:
Procedure: Elective abdominal surgery

SUMMARY:
Worldwide, the rising incidence of obesity has led to the identification of an obesity related syndrome, called metabolic. This syndrome is characterized by central obesity, hypertension, insulin resistance and altered lipid levels.

Taking into consideration the rising incidence of obesity, anesthetists will more frequently encounter patients with metabolic syndrome, in their everyday practice. Moreover, the comorbidities that are related to the metabolic syndrome, increase the risk for perioperative complications. Therefore, strategies that will evaluate and modify the risk will be of great importance in the management of these patients, in order to maximize peri-anaesthetic and surgical safety.

The aim of the study is to assess the incidence of metabolic syndrome and the impact of its presence on the outcome of patients undergoing elective laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients are undergoing elective laparotomy of estimated duration of more than one hour. All operations will be performed under general anesthesia.

Exclusion Criteria:

* Endstage neoplasia
* Procedures performed within 1 hour of admission
* Emergency cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population: Adult patients are undergoing elective laparotomy of estimated duration of more than one hour. All operations will be performed under general anesthesia.
  Group sample sizes of 42 in group one and 42 in group two achieve 90% power to detect a difference between the group proportions of 0,2500. The proportion in group one (MetS group) is assumed to be 0,0500 under the null hypothesis and 0,3000 under the alternative hypothesis. The proportion in group two (the Non-MetS group) is 0,0500. The test statistic used is the two-sided Likelihood Ratio test. The significance level of the test was targeted at 0,0500. The significance level actually achieved by this design is 0,0909.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Perioperative and postoperative adverse cardiac and cerebrovascular events as defined by European Perioperative Clinical Outcome (EPCO) definitions guidelines. | 2 Weeks
Postoperative pulmonary complications as defined by European Perioperative Clinical Outcome (EPCO) definitions guidelines. | 2 Weeks
Acute Kidney Injury (AKI) as defined by Kidney Disease Improving Global Outcomes (KDIGO) guidelines | 2 Weeks
Surgical site infection (superficial or deep) as defined by European Perioperative Clinical Outcome (EPCO) definitions guidelines. | 2 Weeks